CLINICAL TRIAL: NCT05795738
Title: Effects of Different Visual-perceptual-motor Training Courses on Kindergarten Children
Brief Title: Visual Perceptual Motor Training on Kindergarteners
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A-ER-111-161
Record Dates: First submitted 2023-03-05; First posted 2023-04-03 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-05

CONDITIONS: Agraphia
Keywords: Visual; Kindergarten; Chinese
MeSH Terms: conditions — Agraphia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors are blinded to the assigned group of participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): regular kindergarten education
- Chinese characters-based visual-motor program (Experimental): visual perceptual motor activities using Chinese characters as activity materials.
  Interventions: Behavioral: Chinese character-based visuomotor training program
- traditional visual-motor training program (Experimental): visual perceptual motor activities using commercial or self-designed toys and pencil-paper sheets as activity materials.
  Interventions: Behavioral: traditional visuomotor training program

INTERVENTIONS:
Behavioral: Chinese character-based visuomotor training program — this program includes visual-perceptual-motor play, paper-pencil activities, and ipad games using Chinese character as activity materials
  Arms: Chinese characters-based visual-motor program
Behavioral: traditional visuomotor training program — this program includes play and paper-and-pencil activities, ipad games using commercial or self-designed stuffs as activity materials
  Arms: traditional visual-motor training program

SUMMARY:
The study aims to investigate the effects of different visuomotor training programs on children's visuomotor skills and handwriting performance.

DETAILED DESCRIPTION:
The purpose of this project is to investigate the effectiveness of visuomotor activities with different activity materials on fine motor, visual perception, visual-motor integration and handwriting performance of kindergarten children. Kindergarteners will be randomized into the three groups: control, Chinese, and traditional groups. Children in the Chinese and traditional groups will receive a visual perceptual motor training program twice every week for 12 weeks and those in the control group will not receive any intervention during the study period. in the end of fall semester of the first grade, the effectiveness of the interventional programs on handwriting performance of participants will be examined again.

ELIGIBILITY:
Inclusion Criteria:

* Kindergarten children who will study the first grade in coming September
* Both parents are native Mandarin Chinese speakers

Exclusion Criteria:

* A diagnosis of significant neurological, muscular, and skeletal system disorders
* Visual or hearing problems that cannot be corrected to be normal
* Genetic or chromosomal abnormality
* Significant neurological, muscular, and skeletal damage to the trunk or upper extremities
* moderate or severe intellectual disabilities

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The Chinese Handwriting Test | baseline, after 12-week intervention, through study completion, an average of 1 year
  the change of the handwriting performance
The Chinese character recognition Test | baseline, after 12-week intervention, through study completion, an average of 1 year
  the change of the Chinese character recognition ability
The Chinese Handwriting Evaluation Form (preschool version) | baseline, after 12-week intervention
  the change of handwriting performance by kindergarten teacher's rating
The Chinese Handwriting Evaluation Form (School-aged version) | through study completion, an average of 1 year
  the change of handwriting skills by teacher's rating
The Battery of Chinese Basic Literacy | through study completion, an average of 1 year
  the change of reading and handwriting skills

SECONDARY OUTCOMES:
Test of Visual Perceptual Skills-Fourth Edition (TVPS-4) | baseline, after 12-week intervention, through study completion, an average of 1 year
  the change of visual perceptual skills
The Bruininks-Oseretsky Test of Motor Proficiency-Second Edition (BOT-2) | baseline, after 12-week intervention, through study completion, an average of 1 year
  the change of fine motor skills
The Berry-Buktenica Developmental Test of Visual-Motor Integration- Forth Edition (VMI) | baseline, after 12-week intervention, through study completion, an average of 1 year
  the change of VMI

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Shwu Hwang, ScD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD are to be shared with other researchers

REFERENCES:
- [Background] Chen YN, Lin CK, Wei TS, Liu CH, Wuang YP. The effectiveness of multimedia visual perceptual training groups for the preschool children with developmental delay. Res Dev Disabil. 2013 Dec;34(12):4447-54. doi: 10.1016/j.ridd.2013.09.023. Epub 2013 Oct 11. PMID 24120756
- [Background] Chang SH, Yu NY. Visual and Haptic Perception Training to Improve Handwriting Skills in Children With Dysgraphia. Am J Occup Ther. 2017 Mar/Apr;71(2):7102220030p1-7102220030p10. doi: 10.5014/ajot.2017.021311. PMID 28218589
- [Background] Dankert HL, Davies PL, Gavin WJ. Occupational therapy effects on visual-motor skills in preschool children. Am J Occup Ther. 2003 Sep-Oct;57(5):542-9. doi: 10.5014/ajot.57.5.542. PMID 14527116
- [Background] Daly CJ, Kelley GT, Krauss A. Relationship between visual-motor integration and handwriting skills of children in kindergarten: a modified replication study. Am J Occup Ther. 2003 Jul-Aug;57(4):459-62. doi: 10.5014/ajot.57.4.459. PMID 12911088
- [Background] Feder KP, Majnemer A, Bourbonnais D, Platt R, Blayney M, Synnes A. Handwriting performance in preterm children compared with term peers at age 6 to 7 years. Dev Med Child Neurol. 2005 Mar;47(3):163-70. doi: 10.1017/s0012162205000307. PMID 15739720
- [Background] Feder KP, Majnemer A. Handwriting development, competency, and intervention. Dev Med Child Neurol. 2007 Apr;49(4):312-7. doi: 10.1111/j.1469-8749.2007.00312.x. PMID 17376144
- [Background] Hwang YS, Su PF, Hsiao YL, Tsai WH, Hung JY. Developing a Nomogram Model to Predict the Risk of Poor Chinese Handwriting in First Grade. Am J Occup Ther. 2020 Sep/Oct;74(5):7405205080p1-7405205080p8. doi: 10.5014/ajot.2020.038711. PMID 32804626
- [Background] Lee TI, Howe TH, Chen HL, Wang TN. Predicting Handwriting Legibility in Taiwanese Elementary School Children. Am J Occup Ther. 2016 Nov/Dec;70(6):7006220020p1-7006220020p9. doi: 10.5014/ajot.2016.016865. PMID 27767941
- [Background] Ohl AM, Graze H, Weber K, Kenny S, Salvatore C, Wagreich S. Effectiveness of a 10-week tier-1 response to intervention program in improving fine motor and visual-motor skills in general education kindergarten students. Am J Occup Ther. 2013 Sep-Oct;67(5):507-14. doi: 10.5014/ajot.2013.008110. PMID 23968788
- [Background] Poon KW, Li-Tsang CW, Weiss TP, Rosenblum S. The effect of a computerized visual perception and visual-motor integration training program on improving Chinese handwriting of children with handwriting difficulties. Res Dev Disabil. 2010 Nov-Dec;31(6):1552-60. doi: 10.1016/j.ridd.2010.06.001. PMID 20621444
- [Background] Prunty M, Barnett AL, Wilmut K, Plumb M. Visual perceptual and handwriting skills in children with Developmental Coordination Disorder. Hum Mov Sci. 2016 Oct;49:54-65. doi: 10.1016/j.humov.2016.06.003. Epub 2016 Jun 18. PMID 27327259
- [Background] Ratzon NZ, Efraim D, Bart O. A short-term graphomotor program for improving writing readiness skills of first-grade students. Am J Occup Ther. 2007 Jul-Aug;61(4):399-405. doi: 10.5014/ajot.61.4.399. PMID 17685172
- [Background] Taverna L, Tremolada M, Dozza L, Zanin Scaratti R, Ulrike D, Lallo C, Tosetto B. Who Benefits from An Intervention Program on Foundational Skills for Handwriting Addressed to Kindergarten Children and First Graders? Int J Environ Res Public Health. 2020 Mar 24;17(6):2166. doi: 10.3390/ijerph17062166. PMID 32214003
- [Background] Tse LF, Thanapalan KC, Chan CC. Visual-perceptual-kinesthetic inputs on influencing writing performances in children with handwriting difficulties. Res Dev Disabil. 2014 Feb;35(2):340-7. doi: 10.1016/j.ridd.2013.11.013. Epub 2013 Dec 11. PMID 24333804
- [Background] Tseng MH, Chow SM. Perceptual-motor function of school-age children with slow handwriting speed. Am J Occup Ther. 2000 Jan-Feb;54(1):83-8. doi: 10.5014/ajot.54.1.83. PMID 10686631
- [Background] van Hartingsveldt MJ, Cup EH, Hendriks JC, de Vries L, de Groot IJ, Nijhuis-van der Sanden MW. Predictive validity of kindergarten assessments on handwriting readiness. Res Dev Disabil. 2015 Jan;36C:114-124. doi: 10.1016/j.ridd.2014.08.014. Epub 2014 Oct 16. PMID 25462472
- [Background] Volman MJ, van Schendel BM, Jongmans MJ. Handwriting difficulties in primary school children: a search for underlying mechanisms. Am J Occup Ther. 2006 Jul-Aug;60(4):451-60. doi: 10.5014/ajot.60.4.451. PMID 16915876